CLINICAL TRIAL: NCT05826028
Title: Mayzent (Siponimod) Onboarding of Secondary Progressive Multiple Sclerosis (SPMS) Patients With MSGo
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CBAF312AAU02
Record Dates: First submitted 2023-04-19; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Secondary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This study was a retrospective, non-interventional, longitudinal, descriptive study. This study did not have a key underlying hypothesis, rather it was designed to explore the onboarding and adherence of SPMS patients in Australia to Mayzent (siponimod) treatment.

Initiating siponimod involves pre-screen tests, including a CYP2C9 genotype test to determine siponimod maintenance dosing, and patients underwent a 6-day titration prior to maintenance. The MSGo platform was developed to support onboarding. It is an integrated digital platform that functions as a patient support service.

ELIGIBILITY:
Inclusion criteria

* Adult patients with SPMS as per the treating physician's clinical assessment (Therapeutic Goods Administration [TGA]-approved indication of Mayzent).
* Expanded Disability Status Scale (EDSS) of 3.0 to 6.5 (inclusive).
* Patients accessing Mayzent via the Mayzent Experience Program (MEP) must have met the MEP criteria, and if available, the Pharmaceutical Benefits Scheme (PBS) restrictions recommended by the Pharmaceutical Benefits Advisory Committee (PBAC).
* Patients accessing Mayzent via the PBS must have met the PBS restrictions.

Exclusion criteria

* Patients who were contraindicated for Mayzent treatment according to the TGA-approved Product Information.
* Patients diagnosed with clinically isolated syndrome or primary progressive multiple sclerosis (MS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Average time for siponimod onboarding | Up to 168 days

SECONDARY OUTCOMES:
Time to siponimod onboarding in pre-specified sub-groups | Up to 168 days
Percentage of patients who adhered to the titration protocol | Up to 168 days
Time on maintenance therapy | Up to 168 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Australia (2):
  - Novartis Investigational Site, Camperdown, New South Wales
  - Novartis Investigational Site, St Leonards, New South Wales